CLINICAL TRIAL: NCT07380152
Title: Corticosteroid Treatment for Post-COVID-19 Persistent Interstitial Lung Disease
Brief Title: Corticosteroid Therapy in Pulmonary Sequelae of Covid-19
Acronym: COPOSTCOVID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rosangela Villela Garcia, Medical doctor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 47222421.7.0000.5440
Record Dates: First submitted 2024-12-04; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Pulmonary Complications
Keywords: Corticosteroid therapy in post-COVID-19 pulmonary sequelae; post-COVID-19 pulmonary disease; Interstitial lung disease; treatment DPI post-COVID-19
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: The study will be conducted at the Hospital das Clínicas of the Ribeirão Preto School of Medicine of the University of São Paulo. It will be a randomized, double-blind, placebo-controlled study of patients who had pneumonia caused by the novel coronavirus and were treated as outpatients, hospitalized, or who required oxygen therapy or orotracheal intubation.
  After 12 to 20 weeks of the diagnosis of pneumonia caused by the new coronavirus patients will be a standardized time. A medical evaluation, laboratory, imaging, and functional tests will be carried out with a view to immediate entry into the study. This will be considered the first visit. Patients will be randomized, and treatment will be given on the first visit. The evaluations will be carried out on this first visit (baseline) and will be repeated after 3 and 6 months from the first visit. The recruitment period will be 12 months, and the follow-up period for each patient will be 9 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Numbers 1 to 100 were randomly mixed up using a computer randomizer program. The first fifty were allocated as placebo and the last fifty as Treatment. Included patients received a number consecutively from 1 to 100. Only one researcher (EOV) knew to which group every number (patient) belonged, placebo or treatment. This researcher labeled medicine vials accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Treatment: corticosteroid therapy with prednisolone at a dose of half a milligram per kilogram per day, lasting 1 month, which will be gradually withdrawn with a 50% reduction in the dose every 7 days, up to a minimum dose of 5 mg for 7 days before stopping completely. The placebo group will receive tablets identical to prednisolone 20 mg for 1 month, and then the reduction will be done with placebo tablets identical to the 20 mg and 5 mg tablets.
  The identification of the bottles and the preparation of the placebo tablets will be carried out by a compounding pharmacy that will identify the labels by codes, and a researcher on the team will learn the content related to each code (placebo or prednisolone). This researcher will not have access to the study care or procedures.
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Patients who received placebo took a similar number of tablets for similar time span.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Prednisone in anti-inflammatory dose
  Other Names: Corticosteroid therapy

SUMMARY:
Introduction: The new coronavirus (SARS-CoV-2) is a virus with an intense capacity for dissemination and high mortality rate. The main cause of death is viral pneumonia, characterized as organizing pneumonia that responds to treatment with corticosteroids. After 1 month of the acute phase, 25% of patients have complete recovery from lung lesions. However, lung lesions can evolve as persistent interstitial lung disease; it is possible that this persistent disease is also responsive to corticosteroid therapy. There are no controlled and randomized studies on any treatment and its effect on the natural history of this subacute or late manifestation of COVID-19.

Objective: To understand the effect of oral corticosteroid therapy in the treatment of persistent pulmonary manifestations (clinical and radiological) in patients who had moderate, severe, and critical forms of COVID-19. To understand the role of some risk factors in the development of this form of lung disease. To add information on the natural history of interstitial lung disease secondary to SARS-CoV-2 pulmonary infection.

Methodology: Randomized, double-blind, placebo-controlled study of patients who had COVID-19 viral pneumonia. Patients included after 12 weeks of COVID-19 diagnosis with RT-PCR or imaging tests that confirm the infection for inclusion in the protocol 100 patients with changes in high-resolution chest tomography and diffusion spirometry, will be divided into two groups, placebo and treatment; the treatment group will receive prednisolone at a dose of 0.5 mg/kg/day for 1 month and weaning in 30 days. Clinical, laboratory, functional, and imaging evaluations will be performed at the beginning, after 3 and 6 months of treatment and monthly telephone calls.

The evaluation will include a medical evaluation aimed at the cardiopulmonary assessment, arterial blood gas analysis at rest and after 6MWT; functional assessment with spirometry with measurements of FEV1, FVC, TLC, and DLCO; functional assessment during exercise with 6MWT; functionality questionnaires with SF-36, MMRC, and PCFS; and collection of laboratory tests including inflammatory markers - D-dimers, blood count, C-reactive protein and ESR, autoimmunity markers (ANA and RF), and collection of medical and laboratory history data during the acute infection to verify correlation with residual lung disease. Imaging evaluation will be performed with high-resolution chest tomography.

DETAILED DESCRIPTION:
The first case of the new coronavirus (SARS-CoV-2) was recorded in Wuhan, China.

A virus with a high capacity for dissemination, after 4 months, there were already 200,000 deaths caused by COVID-19 worldwide, and high incidence has a high lethality rate.

Up to 20% of affected patients require hospitalization and oxygen therapy, more than 5% of those affected will require intensive care and orotracheal intubation or critical cases, and 2 to 3% will die regardless of the treatment instituted.

The coronavirus infects human cells by binding to the angiotensin-converting enzyme 2 (ACE2) receptor, a receptor present in cells of the lung, heart, kidney, and intestinal tissue (WU et al., 2020).

In lung tissue, it causes damage to the alveolar epithelium, which directly impacts the reduction of the gas exchange area, leading to a decrease in the diffusion capacity of oxygen and carbon dioxide. After the acute phase of the injury, the repair phase of the damaged tissue begins, and the gas exchange area improves, in most cases, enough for the patient to be removed from mechanical ventilation, but there will be extensive lung injury that is still in the recovery phase. At the time, lung tissue injury with characteristics of DAD was already evident, with the presence of multinucleated pneumocytes, which are secondary to the aggression of these cells and proliferation of intrabronchial fibro granular tissue (similar to organizing pneumonia or bronchiolitis obliterans - BOOP) (TSE et al., 2004), evidencing lymphocytic alveolitis, acute fibrinoid injury, and organizing pneumonia (REMMELINK et al., 2020).

In fatal forms, there is DAD with deposition of fibrinous exudate, formation of hyaline membrane, hyperplasia and loss of type 2 pneumocytes, loss of continuity of the basement membrane, and thickening of the alveolar tissue (WIGÉN et al., 2020).

Some people are more susceptible to developing the severe form of coronavirus, such as men, the elderly, diabetics, and obese people. The justification for the worse evolution of the clinical picture for some groups to the detriment of others is that for predisposed people, the severe form of coronavirus has a weaker innate and adaptive response to the action of the virus, which would explain why children and women are less susceptible to the severe pulmonary form (WIGÉN et al., 2020).

After acute lung injury, a process of repair of the alveolar structures begins with stem cells present in the tissue itself. Alveolar macrophages phagocytose the injured tissue, produce cytokines and growth factors involved in tissue repair, and stimulate the differentiation of these cells for the formation of new tissue and deposition of connective tissue. Injury to the pulmonary epithelium and endothelium occurs in the inflammatory phase of COVID-19, as there is dysregulation in the matrix of metalloproteinases (MO et al., 2020)(RAI; SHARMA; KUMAR, 2020). However, when extensive lung injury occurs and the deposition of excess connective tissue and migration of fibroblasts that become myofibroblasts forming fibrotic tissue (OJO et al., 2020). What remains unknown is why certain individuals develop sequelae due to the accumulation of myofibroblasts and excessive collagen deposition, while others recover quickly and completely (RAI; SHARMA; KUMAR, 2020).

The risk factors for the development of persistent interstitial lung disease are related to the greater severity of the disease and are older age, greater severity of lung involvement, increased lactic dehydrogenase (LDH) secondary to the extent of damage to lung tissue in the acute phase of the disease, stay in the intensive care unit, time of orotracheal intubation, smoking and alcoholism (OJO et al., 2020).

Another factor related to the severity of the condition is lymphopenia. The measurement taken at the beginning of the condition predicts a risk of greater lung damage and worse lung recovery since the reduction in lymphocytes causes a deficiency in viral clearance and greater damage to the organism (WIGÉN et al., 2020). The urea level at the beginning of the condition is also related to the aggressiveness of the kidney injury and predicts a worse lung prognosis.

The possible mechanism that would explain persistent lung injuries is that the virus when binding to angiotensin-converting enzyme 2 (ACE2) receptors, internalizes the receptor, and thus, the virus gains access to the cell and begins to attack the organism. Due to downregulation, there is a reduction in the expression of the ACE2 receptor. However, this receptor is part of the renin-angiotensin system, which plays an important role in regulating the immune response and in the recovery of damaged tissue (WIGÉN et al., 2020). Thus, the process of regulating the inflammatory response and recovering lung tissue is impaired, which allows for greater aggression to the lung parenchyma.

There are some differences between the lung disease caused by the new coronavirus and other forms of acute respiratory distress syndrome (ARDS), despite the intense aggression, with lung involvement being the main predictor of severity and sequelae of all of them. COVID-19 has a peculiarity: it causes alveolar damage with low elastance, while others have high elastance. In addition, the computed tomography findings are different from the classic findings of ARDS due to other etiologies, and altered coagulation is also a finding exclusive to COVID-19. In addition to these typical characteristics, residual interstitial lung disease in COVID-19 is different from other fibrosing diseases, such as idiopathic pulmonary fibrosis and fibrosing interstitial lung diseases, as they are mainly marked by the involvement of the pulmonary endothelium, while COVID-19 is marked by the involvement of the alveolar epithelium (RAI; SHARMA; KUMAR, 2020).

Recovery from the pulmonary condition is a slow process, and patients remain symptomatic for a long period, with dyspnea being a very common symptom. Patients who recover, including those with mild symptoms, maintain fatigue in 53% of cases, dyspnea on exertion in 43%, and chest pain in 21.7%, showing that there is a functional pulmonary sequelae in patients who have recovered from COVID-19 (CARFÌ; BERNABEI; LANDI, 2020).

Functional tests to assess possible pulmonary sequelae show that even mild cases can have diffusion changes, and as the severity of the disease increases, the change becomes greater. Functional tests capable of detecting changes are the measurement of carbon monoxide diffusion (DLCO), with an average reduction of 47%, and total lung capacity, with a reduction of 25% after the end of symptoms. These data are even worse in more severe patients (MO et al., 2020), (NUSAIR, 2020). In a 3-month follow-up after hospital discharge, up to 25% of patients maintain diffusion changes (HUANG et al., 2021). Another follow-up study, after 3 months of hospital discharge, showed that up to 25% of patients maintain spirometric changes. And, 9 out of 55 people evaluated (16.3%), even with mild symptoms of the disease in the acute phase, maintained diffusion changes (ZHAO et al., 2020).

Chest computed tomography is the exam that defines the severity of aggression against the lung parenchyma in a quantitative way. Extensive lesions, interstitial thickening, ground-glass opacities, irregular interface, thick reticular pattern, and parenchymal bands predict a greater degree of progression to residual interstitial lung disease.

A study that evaluated lung lesions in the short term after hospital discharge, with serial tomography scans, showed that there was an improvement in lung lesions in 4 weeks in up to 64.7% of patients (consolidations from 49% to 2%, focal ground-glass opacities from 17.7% to 9.8%, multiple ground-glass opacities from 80.4% to 23.5%, interlobular septal thickening from 80.4% to 35.3%, subpleural lines from 29.4% to 7.8%, irregular lines from 41.2% to 15.7%) and disappeared completely in 25.5% of patients (LIU et al., 2020). This shows that most of the changes are inflammatory and largely recover after one month of hospital discharge. However, persistent lesions can progress to persistent interstitial lung disease.

Research project, June 23, 2021 In another study, in patients who required mechanical ventilation, follow-up after 3 months showed complete recovery of lung lesions in only 2 of the 41 patients evaluated. In this study, 89% of patients still had ground-glass opacities according to computed tomography (CT), signs of reticulation and fibrotic bands, with and without parenchymal distortion, bronchiectasis and bronchiolectasis in up to 67% of cases, presence of emphysematous destruction or cavities, with worsening and of pre-existing emphysema. Some patients presented areas of air retention, but this was not a frequent finding, and traction bronchiectasis was rare. This study showed that pulmonary sequelae in patients who had extensive lung involvement are very common and can progress to permanent interstitial lung disease. Also, most people who required mechanical ventilation had changes in lung function and residual changes visualized on high-resolution CT (HRCT) (VAN GASSEL et al., 2021).

The evaluation after 6 months of hospital discharge of patients with COVID-19 showed persistent pulmonary changes on CT in 52% of individuals who did not require oxygen support and 54% of those who required mechanical ventilation, noninvasive ventilation, or other ventilatory support. Regarding DLCO, even patients with the mild form of the disease may maintain alterations, present in 22% of patients who did not require oxygen therapy and in 56% of patients who required some type of ventilatory support (HUANG et al., 2021).

The treatment of the pulmonary condition still in the acute phase in patients requiring orotracheal intubation and oxygen therapy (DE BACKER; AZOULAY; VINCENT, 2020) demonstrated benefit with immunosuppressive doses of corticosteroid therapy due to a pattern of injury to the lung tissue with lymphocytic alveolitis, acute fibrinoid injury and organizing pneumonia (REMMELINK et al., 2020), all of which are acute alterations responsive to corticosteroid therapy.

In hospitalized patients, the use of corticosteroid therapy with dexamethasone and methylprednisolone has the potential to reduce mortality. Furthermore, the comparison between the two types of corticosteroids showed that the use of methylprednisolone was more effective (KO et al., 2021).

After the recovery period, interstitial lung disease persists in many patients, but the lesions are not characteristic of definitive fibrosis with honeycombing. According to RAI et al., 2020 (RAI; SHARMA; KUMAR, 2020), the studies reviewed in the literature designated the pulmonary sequelae as pulmonary fibrosis. However, in a recent study, it was called persistent interstitial lung involvement due to the lack of definitive characteristics of a fibrosing lesion and the presence of possible reversible lesions (WELLS; DEVARAJ; DESAI, 2021).

The evaluation time to confirm persistent lung disease and the period of natural recovery from the disease are still uncertain. However, data from the literature on the follow-up of severe pneumonia show that the radiological recovery time should be around six weeks. Regarding MERS and SARS-CoV-1, the radiological recovery time is around 12 weeks, with complete resolution of radiological alterations in two-thirds of patients during this period, and the maintenance of radiological alterations after this period indicates a high probability of permanent lung disease (GEORGE et al., 2020). This review also suggests a post-COVID-19 follow-up after 12 weeks with chest X-ray, diffusion measurements, and walk test to assess desaturation during exertion, and if any alteration is identified, a chest HRCT scan is considered to assess interstitial lung disease. However, the initial assessment or screening performed only with a simple chest X-ray may lead to the non-identification of pulmonary sequelae due to its low sensitivity.

Follow-up of patients after 6 months of hospital discharge showed changes in chest X-rays in up to 25% of patients and reduced diffusion in 46%, but only 31% of patients had dyspnea on exertion with MMRC greater than or equal to 1 (FAVERIO et al., 2021), the most severe patients are those with greater impairment in diffusion capacity and changes in imaging tests (HUANG et al., 2021).

Studies on which treatment would be most effective for persistent interstitial disease have not yet been established in the medical literature, and the medications currently being tested are nintedanib, pirfenidone, chloroquine, and corticosteroids. Prophylactic measures such as protective mechanical ventilation techniques, measures to prevent pneumonia infections and other respiratory complications can reduce the risk of residual lung disease (RAI; SHARMA; KUMAR, 2020).

A study on the use of corticosteroids in patients with pulmonary sequelae showed significant improvement after the use of a dose of 0.5 mg/kg, but with rapid weaning and weaning beginning in the first week of use. This study did not have a control group, and patients were followed for 3 months only after inclusion and initiation of treatment (MYALL et al., 2021). The use of corticosteroids plays a crucial role in the treatment of inflammatory lung disease related to COVID-19, apparently in all phases of the disease.

Since COVID-19-related lung lesions in the acute phase are responsive to corticosteroid therapy, it is inferred that, for persistent interstitial lung disease that demonstrates an inflammatory pattern with alveolar involvement, corticosteroid therapy may also have an important role. There are no controlled and randomized studies on any treatment and its effect on the natural history of this complication of COVID-19.

ELIGIBILITY:
Inclusion criteria

* Over 18 years of age;
* Diagnosis of COVID-19 by RT-PCR (Reverse transcription polymerase chain reaction), a test that detects the presence of viral antigen in nasal and oropharyngeal secretions or chest tomography typical of COVID-19 according to radiological standardization for COVID-19 cases (Machnicki, 2021);
* Pulmonary involvement with persistent disease identified on high-resolution computed tomography of the chest;
* Reduction in DLCO (percentage of predicted), with measurements less than or equal to 80%.

Exclusion criteria

* Previous diagnosis of pulmonary embolism;
* Previous and decompensated heart failure with electrocardiographic changes, chest X-ray with increased cardiac silhouette, and signs in the clinical examination suggestive of heart failure;
* History of acute myocardial infarction in the last month or angina pectoris; Absolute contraindications to the use of corticosteroids or other comorbidities that prevent the use of corticosteroids such as uncontrolled diabetes, untreated glaucoma, current infections such as pneumonia or tuberculosis, and untreated psychiatric disorders;
* Pregnancy and lactation;
* Inability to perform stress tests such as walking tests and spirometry due to critically ill neuropathy or sequelae of stroke, among other limiting pathologies.

The patient will be informed of the risks related to corticosteroid treatment, and this information will be included in the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
The rate of radiological, functional and quality of life improvement in prednisolone treatment for persistent interstitial lung disease following SARS-CoV-2. | 10 months
  Rate of improvement, after treatment with prednisolone, of radiological, functional, and quality of life parameters in patients with persistent interstitial lung disease resulting from SARS-CoV-2 infection, in moderate, severe, and critical forms of COVID-19. Assessments were performed at 4, 7, and 10 months after diagnosis, .

SECONDARY OUTCOMES:
The incidence of risk factors that may influence the severe outcome of COVID-19 lung disease. | In the first evaluation, 4 months after diagnosis.
  The incidence of some risk factors in the development of this form of lung disease.
Monitoring of post-COVID lung disease. | During recruitment and monitoring.
  To add information on the natural history of interstitial lung disease secondary to SARS-CoV-2 pulmonary infection.

CONTACTS AND LOCATIONS:
Overall Officials: Elcio O. Vianna, Professor, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Due to the confidentiality of the double-blind study and the protection of patient data, the study has not yet been published. The data will be sent to the journal in which the publication will be made.

REFERENCES:
- [Background] Zhao YM, Shang YM, Song WB, Li QQ, Xie H, Xu QF, Jia JL, Li LM, Mao HL, Zhou XM, Luo H, Gao YF, Xu AG. Follow-up study of the pulmonary function and related physiological characteristics of COVID-19 survivors three months after recovery. EClinicalMedicine. 2020 Aug;25:100463. doi: 10.1016/j.eclinm.2020.100463. Epub 2020 Jul 15. PMID 32838236
- [Background] Wu F, Zhao S, Yu B, et al. Complete genome characterisation of a novel coronavirus associated with severe human respiratory disease in Wuhan, China. bioRxiv; 2020. DOI: 10.1101/2020.01.24.919183.
- [Background] Wigen J, Lofdahl A, Bjermer L, Elowsson-Rendin L, Westergren-Thorsson G. Converging pathways in pulmonary fibrosis and Covid-19 - The fibrotic link to disease severity. Respir Med X. 2020 Nov;2:100023. doi: 10.1016/j.yrmex.2020.100023. Epub 2020 Oct 9. PMID 33083782
- [Background] Wells AU, Devaraj A, Desai SR. Interstitial Lung Disease after COVID-19 Infection: A Catalog of Uncertainties. Radiology. 2021 Apr;299(1):E216-E218. doi: 10.1148/radiol.2021204482. Epub 2021 Jan 26. No abstract available. PMID 33502279
- [Background] van Gassel RJJ, Bels JLM, Raafs A, van Bussel BCT, van de Poll MCG, Simons SO, van der Meer LWL, Gietema HA, Posthuma R, van Santen S. High Prevalence of Pulmonary Sequelae at 3 Months after Hospital Discharge in Mechanically Ventilated Survivors of COVID-19. Am J Respir Crit Care Med. 2021 Feb 1;203(3):371-374. doi: 10.1164/rccm.202010-3823LE. No abstract available. PMID 33326353
- [Background] Tse GM, To KF, Chan PK, Lo AW, Ng KC, Wu A, Lee N, Wong HC, Mak SM, Chan KF, Hui DS, Sung JJ, Ng HK. Pulmonary pathological features in coronavirus associated severe acute respiratory syndrome (SARS). J Clin Pathol. 2004 Mar;57(3):260-5. doi: 10.1136/jcp.2003.013276. PMID 14990596
- [Background] Remmelink M, De Mendonca R, D'Haene N, De Clercq S, Verocq C, Lebrun L, Lavis P, Racu ML, Trepant AL, Maris C, Rorive S, Goffard JC, De Witte O, Peluso L, Vincent JL, Decaestecker C, Taccone FS, Salmon I. Unspecific post-mortem findings despite multiorgan viral spread in COVID-19 patients. Crit Care. 2020 Aug 12;24(1):495. doi: 10.1186/s13054-020-03218-5. PMID 32787909
- [Background] Rai DK, Sharma P, Kumar R. Post covid 19 pulmonary fibrosis. Is it real threat? Indian J Tuberc. 2021 Jul;68(3):330-333. doi: 10.1016/j.ijtb.2020.11.003. Epub 2020 Nov 10. PMID 34099197
- [Background] Ojo AS, Balogun SA, Williams OT, Ojo OS. Pulmonary Fibrosis in COVID-19 Survivors: Predictive Factors and Risk Reduction Strategies. Pulm Med. 2020 Aug 10;2020:6175964. doi: 10.1155/2020/6175964. eCollection 2020. PMID 32850151
- [Background] Nusair S. Abnormal carbon monoxide diffusion capacity in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jul 23;56(1):2001832. doi: 10.1183/13993003.01832-2020. Print 2020 Jul. PMID 32703822
- [Background] Myall KJ, Mukherjee B, Castanheira AM, Lam JL, Benedetti G, Mak SM, Preston R, Thillai M, Dewar A, Molyneaux PL, West AG. Persistent Post-COVID-19 Interstitial Lung Disease. An Observational Study of Corticosteroid Treatment. Ann Am Thorac Soc. 2021 May;18(5):799-806. doi: 10.1513/AnnalsATS.202008-1002OC. PMID 33433263
- [Background] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Liu C, Ye L, Xia R, Zheng X, Yuan C, Wang Z, Lin R, Shi D, Gao Y, Yao J, Sun Q, Wang X, Jin M. Chest Computed Tomography and Clinical Follow-Up of Discharged Patients with COVID-19 in Wenzhou City, Zhejiang, China. Ann Am Thorac Soc. 2020 Oct;17(10):1231-1237. doi: 10.1513/AnnalsATS.202004-324OC. PMID 32692945
- [Background] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Background] Ko JJ, Wu C, Mehta N, Wald-Dickler N, Yang W, Qiao R. A Comparison of Methylprednisolone and Dexamethasone in Intensive Care Patients With COVID-19. J Intensive Care Med. 2021 Jun;36(6):673-680. doi: 10.1177/0885066621994057. Epub 2021 Feb 25. PMID 33632000
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306
- [Background] The Lancet Editors. Retraction and republication: 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2023 Jun 17;401(10393):2025. doi: 10.1016/S0140-6736(23)01175-3. Epub 2023 Jun 9. No abstract available. PMID 37307841
- [Background] George PM, Barratt SL, Condliffe R, Desai SR, Devaraj A, Forrest I, Gibbons MA, Hart N, Jenkins RG, McAuley DF, Patel BV, Thwaite E, Spencer LG. Respiratory follow-up of patients with COVID-19 pneumonia. Thorax. 2020 Nov;75(11):1009-1016. doi: 10.1136/thoraxjnl-2020-215314. Epub 2020 Aug 24. PMID 32839287
- [Background] Faverio P, Luppi F, Rebora P, Busnelli S, Stainer A, Catalano M, Parachini L, Monzani A, Galimberti S, Bini F, Bodini BD, Betti M, De Giacomi F, Scarpazza P, Oggionni E, Scartabellati A, Bilucaglia L, Ceruti P, Modina D, Harari S, Caminati A, Valsecchi MG, Bellani G, Foti G, Pesci A. Six-Month Pulmonary Impairment after Severe COVID-19: A Prospective, Multicentre Follow-Up Study. Respiration. 2021;100(11):1078-1087. doi: 10.1159/000518141. Epub 2021 Aug 19. PMID 34515212
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Tradução para a língua portuguesa e validação do questionário genérico de avaliação de qualidade de vida SF-36 (Brasil SF-36) / Brazilian-Portuguese version of the SF-36. A reliable and valid quality of life outcome measure Ciconelli, Rozana Mesquita; Ferraz, Marcos Bosi; Santos, Wilton; Meinão, Ivone; Quaresma, Marina Rodrigues. Rev. bras. reumatol ; Rev. bras. reumatol;39(3): 143-50, maio-jun. 1999.
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Britto RR, Probst VS, de Andrade AF, Samora GA, Hernandes NA, Marinho PE, Karsten M, Pitta F, Parreira VF. Reference equations for the six-minute walk distance based on a Brazilian multicenter study. Braz J Phys Ther. 2013 Nov-Dec;17(6):556-63. doi: 10.1590/S1413-35552012005000122. Epub 2013 Nov 14. PMID 24271092
- [Background] Borg G. Psychophysical scaling with applications in physical work and the perception of exertion. Scand J Work Environ Health. 1990;16 Suppl 1:55-8. doi: 10.5271/sjweh.1815. PMID 2345867
- See also: Tradução para a língua portuguesa e validação do questionário genérico de avaliação de qualidade de vida SF-36 (Brasil SF-36) / Brazilian-Portuguese version of the SF-36. A reliable and valid quality of life outcome measure — https://pesquisa.bvsalud.org/portal/resource/pt/lil-296502
- Available data/document: Individual Participant Data Set: Initial letters of participant — https://redcapbrasil.com.br/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT07380152/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT07380152/ICF_001.pdf